CLINICAL TRIAL: NCT02836262
Title: A Multi-Center Prospective Study of the Hip Innovation Technology (HIT) Hip Replacement System in Primary Total Hip Arthroplasty
Brief Title: Hip Replacement System (HRS-P) in Primary Total Hip Arthroplasty
Acronym: (HRS-P)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hip Innovation Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIT-001
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis of Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIT Hip Replacement System (HRS) (Experimental): Single group assignment with historical controls.
  Interventions: Device: HIT Hip Replacement System

INTERVENTIONS:
Device: HIT Hip Replacement System — HIT Hip Replacement System

SUMMARY:
To evaluate effectiveness and safety of HHRS in subjects undergoing total hip arthroplasty (THA). Effectiveness will be evaluated using patient-reported, clinical, radiologic, and radiostereometric outcomes. Safety will be evaluated through the collection of device-related and unanticipated device-related adverse events.

DETAILED DESCRIPTION:
The HIT Hip Replacement System (HHRS) is a Metal-on-Polyethylene (MoP) conventional hip prosthesis. The HHRS consists of a femoral stem, an acetabular cup and a Cobalt Chromium Molybdenum (CoCrMo) ball that articulates within a polyethylene liner. The ball sits on the acetabular cup, and the polyethylene liner is attached to the femoral cup, which attaches to the femoral stem, instead of the acetabular cup. The acetabular component of the HHRS consists of a hemispherical acetabular shell with a clustered screw-hole design. The outside of the shells are coated with titanium plasma to facilitate bone in-growth and provide secure intermediate fixation with the prepared bone surface at the site of implantation. The acetabular cup has a 3-hole design that accommodates three titanium alloy bone screws. Inside the acetabular cup is a male taper for assembly with the acetabular ball. The femoral component consists of a femoral stem manufactured from titanium and a mating cobalt chrome femoral cup lined with a highly cross-linked ultra-high-molecular-weight polyethylene (UHMWPE). As with the acetabular cup, the femoral stem is porous coated using a plasma spray of pure titanium, which is intended to facilitate bone in-growth and provide secure intermediate fixation with the prepared bone surface at the site of implantation. The femoral stem incorporates a female taper for assembly with the male taper of the femoral cup.

The device has undergone extensive pre-clinical testing. There is no clinical experience with the HRS.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a non-inflammatory degenerative joint disease (NIDJD) or any of its composite diagnoses such as osteoarthritis, avascular necrosis, traumatic arthritis, slipped capital epiphysis, fracture of the pelvis, and diastrophic variant requiring unilateral primary total hip replacement.
* Age between 65 and 79 years (inclusive) at the time of enrollment.
* Patient is a suitable candidate for primary total hip replacement at the discretion of the Investigator.
* Pre-surgery (within 28 days before surgery) WOMAC Global Score of 40 or larger on a scale from 0 (best) to 96 (worst)
* Signed and dated informed consent document.
* Patient is willing and able to participate in required follow-up visits at the Investigational site and to complete study procedures and questionnaires.

Exclusion Criteria:

* Patient has had total hip replacement, hemi-arthroplasty, or fusion in either hip in the last 12 months;
* Patient has planned total hip arthroplasty on a contra-lateral joint in the next 12 months;
* Patient has a known allergy to any component of the study device;
* Patient has a history of active sepsis in the joint;
* Patient has an insufficient acetabular or femoral bone stock in which good anchorage of the implants are unlikely or impossible;
* Patient has total or partial absence of the muscular or ligamentous apparatus;
* Patient has known moderate to severe renal insufficiency;
* Patient has vascular insufficiency, muscular atrophy, or neuromuscular disease in either leg (based on the Investigator's discretion);
* Patient has a deformity of the affected limb or significant anatomic variance of the affected hip;
* Patient has an active malignancy or history of invasive malignancy within the last five years, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated. Patients with carcinoma in situ of the uterine cervix definitively treated more than 1 year prior to enrollment may enter the study;
* Patient has any condition which may, in the opinion of the Investigator, interfere with the total hip replacement survival or patient outcomes (e.g. Paget's disease, Charcot's disease);
* Patient has rheumatoid arthritis or other autoimmune condition that affect joints (e.g. Lupus Arthritis);
* Patient has any condition that would interfere with patient self-assessment or pain, the function or quality of life required for patient reported outcomes during the study (based on the Investigator's discretion);
* Body Mass Index (BMI) of 40 or more;
* Patient has an active infection (e.g. hepatitis, AIDS, ARC) - systemic or at the site of intended surgery;
* Patient is currently participating in any investigational study not related to this study's pre-operative or post-operative care;
* Patient has any other severe acute or chronic medical condition that may interfere with the interpretation of the study results, in the judgment of the Investigator, which would make the patient inappropriate for entry into this study;
* Patient has a history of metabolic bone disease (e.g. Paget's disease or osteomalacia);
* Patient is currently pregnant or is planning to become pregnant.

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-25 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) v3.0 Likert Scale Functional Limitations Score between baseline (pre-operative) and the 730- day post-operative follow-up time point. | between pre-operative and 730 days (24 months)
Change in Harris Hip Score between baseline (pre-operative) and the 730-day post-operative follow-up time point. | between pre-operative and 730 days (24 months)

SECONDARY OUTCOMES:
Change in Oxford Hip Score between 730-day post-operative and baseline (pre-surgery) | between 730-days post-operative and baseline (pre-surgery)
Change in Short Form 36 v2 Physical Component Score (PCS) between 730-days post-operative and baseline (pre-surgery) | between 730-days post-operative and baseline (pre-surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, MD, Principal Investigator — Orthopaedic Innovation Centre; Branko Kopjar, MD, PhD, Study Director — Nor Consult, LLC
Locations (1):
- Orthopaedic Innovation Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No